CLINICAL TRIAL: NCT03306056
Title: Comparison of the Effects of Whole-body Electromyostimulation Versus Conventional Low-volume Strength Training in Overweight Individuals at Increased Cardiometabolic Risk
Brief Title: Whole-body Electromyostimulation Versus Conventional Low-volume Strength Training in Overweight Individuals
Acronym: EKAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EKAM-Study
Record Dates: First submitted 2017-09-27; First posted 2017-10-10 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Overweight and Obesity; Metabolic Syndrome
Keywords: Exercise; Strength Training; Health Promotion; Inflammation; Body Composition
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Motor Activity; Inflammation

STUDY DESIGN:
Intervention Model Description: parallel-group, randomized-controlled study
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessors involved in data analysis will not be aware of the arm to which the participants were allocated (single-blinded masking).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Experimental): Nutritional therapy / no exercise
  Interventions: Other: Control
- Standard Strength Training (Experimental): Nutritional therapy combined with a Standard Strength Training program
  Interventions: Other: Standard Strength Training
- Low-volume Strength Training (Experimental): Nutritional therapy combined with a low-volume Strength Training program
  Interventions: Other: Low-volume Strength Training
- Whole-body Electromyostimulation (Experimental): Nutritional therapy combined with Whole-Body Electromyostimulation
  Interventions: Other: Whole-Body Electromyostimulation (WB-EMS)

INTERVENTIONS:
Other: Control — Individualized, weight-reducing nutritional therapy and counseling, during a study period of 12 weeks
  Arms: Control
Other: Standard Strength Training — Procedures: Nutritional therapy (individualized, weight-reducing nutritional therapy and counseling) during a study period of 12 weeks combined with a standard strength training program:
  * 5 strength training exercises (chest, upper/lower back, abdominals, legs)
  * 3 sets per exercise
  * time-effort per session: ~90 min
  * 2 training sessions per week
  * duration of exercise intervention: 12 weeks
  Arms: Standard Strength Training
Other: Low-volume Strength Training — Procedures: Nutritional therapy (individualized, weight-reducing nutritional therapy and counseling) during a study period of 12 weeks combined a low-volume strength training program:
  * 5 strength training exercises (chest, upper/lower back, abdominals, legs)
  * 1 set per exercise
  * time-effort per session: ~20 min
  * 2 training sessions per week
  * duration of exercise intervention: 12 weeks
  Arms: Low-volume Strength Training
Other: Whole-Body Electromyostimulation (WB-EMS) — Procedures: Nutritional therapy (individualized, weight-reducing nutritional therapy and counseling) during a study period of 12 weeks combined with WB-EMS:
  * time-effort per session: ~20 min
  * duration of exercise intervention: 12 weeks
  Arms: Whole-body Electromyostimulation

SUMMARY:
The main purpose of this study is to compare the effects of whole-body electromyostimulation versus a conventional low-volume strength-training program, each combined with an individualized, weight-reducing diet, on the cardiometabolic risk profile, muscle strength, body composition, inflammatory markers and subjective health outcomes in overweight individuals at increased cardiometabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index >25
* presence of at least 2 cardiometabolic risk factors

Exclusion Criteria:

* Healthy persons or patients under age
* Overweight persons without any additional cardiometabolic risk factors
* Pregnancy, Lactation
* Psychological disorders, epilepsy, sever neurological disorders
* Participation in other exercise- or nutrition studies within the last 6 months
* acute cardiovascular disease
* malignant disease
* Rheuma
* Intake of anabolic drugs,
* Skin injuries in the area of electrode placements
* Electronic implants (defibrillator, pacemaker)
* Persons in mental hospitals by order of authorities or jurisdiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Metabolic Syndrome Z-Score (MetS-Z-Score) | 12 weeks (baseline to 12 week follow-up assessment)
  MetS-Z-Score will be calculated from each individual's measures of waist circumference, mean arterial blood pressure, triglycerides, and HDL-cholesterol, based on equations specific to sex.

SECONDARY OUTCOMES:
Muscle strength | 12 weeks (baseline to 12 week follow-up assessment)
  Muscle strength of the five major muscle groups (chest, upper back, lower back, abdominals, legs) will be assessed by using specific strength-training devices (Butterfly, Pull-down, Hyperextension, Abdominal Crunch, Leg-Press)
Body Composition | 12 weeks (baseline to 12 week follow-up assessment)
  Muscle mass, fat mass and body water will be measured by Bioelectrical Impedance Analysis (BIA)
Cardiorespiratory Fitness (CRF) | 12 weeks (baseline to 12 week follow-up assessment)
  CRF will be assessed by measuring Maximum Oxygen uptake (VO2max)
Inflammation status | 12 weeks (baseline to 12 week follow-up assessment)
  Inflammation will be assessed by measuring Levels of CRP and inflammatory cytokines and other inflammatory blood markers
Health-related quality of life | 12 weeks (baseline to 12 week follow-up assessment)
  Health-related quality of life will be assessed by using the standardized and validated EQ-5D-5L Questionnaire
Pain scores | 12 weeks (baseline to 12 week follow-up assessment)
  Pain scores will be assessed by using the standardized and validated Chronic Pain Grade Questionnaire (CPGQ)
Perceived stress | 12 weeks (baseline to 12 week follow-up assessment)
  Perceived stress will be assessed by using the standardized and validated Perceived Stress Questionnaire (PSQ)
Subjective work ability | 12 weeks (baseline to 12 week follow-up assessment)
  Subjective work ability will be assessed by using the standardized and validated Work Ability Index Questionnaire (WAI)

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Reljic, Dr., Principal Investigator — University Erlangen Nuremberg Medical School; Yurdaguel Zopf, Prof., Principal Investigator — University Erlangen Nuremberg Medical School
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports,, Erlangen, Germany